CLINICAL TRIAL: NCT01934751
Title: Randomized Controlled Trial on the Effectiveness of Immediate Versus Delayed Access to Hospital-based Addiction Services
Brief Title: Effectiveness of a Hospital Addiction Service in Treating Opioid and Alcohol Addiction
Acronym: H-SOAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women's College Hospital (Other)
Collaborators: Unity Health Toronto (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Meldon Kahan, Medical director, Substance Use Service, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRIDGES; MOHLTC (Other: University of Toronto, Ontario Ministry of Health)
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Alcohol Addiction; Opiate Addiction
MeSH Terms: conditions — Alcoholism; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opioid dependent (Other): Subjects with a possible opioid use disorder, as determined by positive responses on the eligibility form: has used opioids within the past 30 days, opioid use has been a problem, and at least one harmful consequence of opioid use has been present (eg. withdrawal symptoms, or problems with family, friends, work, money etc.).
  Interventions: Other: Delayed Intervention (DI); Other: Rapid Intervention (RI)
- Alcohol dependent (Other): Patients who indicate they have a problem with alcohol will be asked to complete the AUDIT, a validated, 10-item instrument that measures the severity of an alcohol problem. The AUDIT enquires about core features of alcohol dependence, such as failure to fulfill obligations. A score of 8 or more indicates possible alcohol dependence.
  Interventions: Other: Delayed Intervention (DI); Other: Rapid Intervention (RI)

INTERVENTIONS:
Other: Delayed Intervention (DI) — Subjects randomized to the DI group will be given a card with the number for the usual Substance Use Service, where they will be seen within 2-4 weeks (standard practice). If they attend the Substance Use Service they will be offered supportive counseling, pharmacotherapy, and information on community treatment resources.
Other: Rapid Intervention (RI) — Subjects randomized to the RI group will be seen in the Substance Use Service at within 1-2 days of study enrolment. The Research Assistant will book the appointment and arrange transportation. At the Substance Use Service they will be offered supportive counseling, pharmacotherapy, and information on community treatment resources.

SUMMARY:
Hypothesis: Patients who are addicted to opioids or alcohol will have reduced substance use, health care utilization if they have immediate and convenient access to pharmacotherapy and addiction counselling.

Summary: This randomized trial will compare two different interventions for 124 alcohol and opioid-addicted patients admitted to either Women's Own Detox (WOD) at the University Health Network or the Withdrawal Management Service (WMS) at Saint Michael's Hospital (SMH. The Delayed Intervention group will receive a card with contact information for the St. Michael's Hospital and Women's College Hospital addiction medicine services. The Rapid Intervention group will be seen by an addiction physician from one of these services, within a day or two of their admission to the WOD or the SMH WMS. The addiction physician will prescribe buprenorphine or anti-alcohol medications, and the physician, nurse and/or therapist will provide ongoing counseling, follow-up and shared care with the family physician. Outcomes (measured at 6 and 12 months) include treatment retention, health care utilization and cost, medications prescribed, and alcohol and opioid use.

ELIGIBILITY:
Inclusion Criteria:

* a possible alcohol use disorder, as determined by a score of 8 or above on the AUDIT (Alcohol Use Disorders Identification Test); or, a possible opioid use disorder, as determined by positive responses on the eligibility form: within the past 30 days, opioid use has been a problem, and at least one harmful consequence of opioid use has been present, eg withdrawal symptoms, or problems with family, friends, work, money etc. If the addiction physician who assesses the patient at the first visit to the addiction service concludes that these screening tests were falsely positive and the patient does not have an alcohol or opioid use disorder, the physician will contact the RA to discharge the patient from the study.
* Interested in receiving treatment at an addiction medicine service.
* is alert and able to provide informed consent (ie is not confused, agitated, hostile, intoxicated, sedated or in severe withdrawal)
* Has attended a hospital Emergency Department or has been admitted to hospital in Ontario within the past year.
* Can speak and read English.

Exclusion Criteria:

* Pregnant
* Currently receiving methadone or buprenorphine treatment
* Cognitively impaired
* Unable to speak or read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Treatment retention | 12 months
  The number of subjects in each group that attend the addiction service, and the mean number of visits per subject.
Healthcare utilization and cost | 36 months
  For each subject the ICES (Institute for Clinical Evaluative Sciences) linked administrative databases will be used to track, from 24 months before to 12 months after the initial visit: a) the number of hospitalizations and number of hospital days (Canadian Institute for Health Information (CIHI) Discharge Abstract Database), b) Emergency Department (ED) visits (CIHI National Ambulatory Care Reporting System), c) primary care visits and outpatient laboratory services (Ontario Health Information Plan Database). During the monthly telephone calls and at the 6 and 12 month visits, the Research Assistant (RA) will ask subjects about recent ED visits, hospitalizations and outpatient medical visits
Prescriptions | 36 months
  For patients eligible for pharmacotherapy, ICES will be used to evaluate pre-post (prescribing from 24 months before study entry to 12 months after) changes in opioid and benzodiazepine prescribing, and prescribing of buprenorphine, methadone, and anti-alcohol drugs.
Substance use | 12 months
  The research assistant will conduct interviews at baseline, 6, and 12 months during which subjects will be asked about changes in substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Meldon Kahan, MDCCFP FRCPC, Principal Investigator — Women's College Hospital; Anita Srivastava, MD MSc CCFP, Principal Investigator — St. Joseph's Health Centre Toronto; Rajesh Gupta, MD MEd FRCPC, Principal Investigator — Unity Health Toronto; Leslie Buckley, MD, MPH, Principal Investigator — University Health Network, Toronto
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Shield, K. D., T. Kehoe, B. Taylor, J. Patra and J. Rehm (2011).
- [Background] Taylor B, Rehm J, Patra J, Popova S, Baliunas D. Alcohol-attributable morbidity and resulting health care costs in Canada in 2002: recommendations for policy and prevention. J Stud Alcohol Drugs. 2007 Jan;68(1):36-47. doi: 10.15288/jsad.2007.68.36. PMID 17149516
- [Background] Center for Disease Control.
- [Background] Dhalla IA, Mamdani MM, Sivilotti ML, Kopp A, Qureshi O, Juurlink DN. Prescribing of opioid analgesics and related mortality before and after the introduction of long-acting oxycodone. CMAJ. 2009 Dec 8;181(12):891-6. doi: 10.1503/cmaj.090784. Epub 2009 Dec 7. PMID 19969578
- [Background] Domingo A, Anto JM, Cami J. Epidemiological surveillance of opioid-related episodes in an emergency room of Barcelona, Spain (1979-1989). Br J Addict. 1991 Nov;86(11):1459-66. doi: 10.1111/j.1360-0443.1991.tb01731.x. PMID 1777740
- [Background] Perez Gonzalez K, Domingo-Salvany A, Hartnoll R. [The characteristics of opiate users seen in an emergency service]. Gac Sanit. 1999 Mar-Apr;13(2):88-95. doi: 10.1016/s0213-9111(99)71332-4. Spanish. PMID 10354528
- [Background] Gowing, L., R. Ali and J. M. White (2009).
- [Background] Hoffman, K. A., J. H. Ford, C. J. Tillotson, D. Choi and D. McCarty (2011).
- [Background] Aszalos R, McDuff DR, Weintraub E, Montoya I, Schwartz R. Engaging hospitalized heroin-dependent patients into substance abuse treatment. J Subst Abuse Treat. 1999 Jul-Sep;17(1-2):149-58. doi: 10.1016/s0740-5472(98)00075-0. PMID 10435263
- [Background] Shanahan CW, Beers D, Alford DP, Brigandi E, Samet JH. A transitional opioid program to engage hospitalized drug users. J Gen Intern Med. 2010 Aug;25(8):803-8. doi: 10.1007/s11606-010-1311-3. Epub 2010 Mar 17. PMID 20237960
- [Background] Miller, P. M., S. W. Book and S. H. Stewart (2011).
- [Background] Fleming MF, Mundt MP, French MT, Manwell LB, Stauffacher EA, Barry KL. Benefit-cost analysis of brief physician advice with problem drinkers in primary care settings. Med Care. 2000 Jan;38(1):7-18. doi: 10.1097/00005650-200001000-00003. PMID 10630716
- [Background] Alford DP, LaBelle CT, Kretsch N, Bergeron A, Winter M, Botticelli M, Samet JH. Collaborative care of opioid-addicted patients in primary care using buprenorphine: five-year experience. Arch Intern Med. 2011 Mar 14;171(5):425-31. doi: 10.1001/archinternmed.2010.541. PMID 21403039
- [Background] Soeffing JM, Martin LD, Fingerhood MI, Jasinski DR, Rastegar DA. Buprenorphine maintenance treatment in a primary care setting: outcomes at 1 year. J Subst Abuse Treat. 2009 Dec;37(4):426-30. doi: 10.1016/j.jsat.2009.05.003. Epub 2009 Jun 23. PMID 19553061
- [Background] Mark TL, Montejano LB, Kranzler HR, Chalk M, Gastfriend DR. Comparison of healthcare utilization among patients treated with alcoholism medications. Am J Manag Care. 2010;16(12):879-88. PMID 21348558
- [Background] McCarty, D., N. A. Perrin, C. A. Green, M. R. Polen, M. C. Leo and F. Lynch (2010).
- [Background] Moreno MA, Vanderstoep A, Parks MR, Zimmerman FJ, Kurth A, Christakis DA. Reducing at-risk adolescents' display of risk behavior on a social networking web site: a randomized controlled pilot intervention trial. Arch Pediatr Adolesc Med. 2009 Jan;163(1):35-41. doi: 10.1001/archpediatrics.2008.502. PMID 19124701
- [Background] Neighbors, C. J., N. P. Barnett, D. J. Rohsenow, S. M. Colby and P. M. Monti
- [Background] Owens L, Butcher G, Gilmore I, Kolamunnage-Dona R, Oyee J, Perkins L, Walley T, Williamson P, Wilson K, Pirmohamed M. A randomised controlled trial of extended brief intervention for alcohol dependent patients in an acute hospital setting (ADPAC). BMC Public Health. 2011 Jul 4;11:528. doi: 10.1186/1471-2458-11-528. PMID 21726445
- [Background] D'Onofrio, G. and L. C. Degutis (2010).
- [Background] Soderstrom CA, DiClemente CC, Dischinger PC, Hebel JR, McDuff DR, Auman KM, Kufera JA. A controlled trial of brief intervention versus brief advice for at-risk drinking trauma center patients. J Trauma. 2007 May;62(5):1102-11; discussion 1111-2. doi: 10.1097/TA.0b013e31804bdb26. PMID 17495708
- [Background] Internet sample size calculator. Hedwig.mgh.harvard.edu. Schoenfield D. statistical considerations for clinical trials and scientific experiments.
- [Background] Kahan M, Wilson L, Midmer D, Ordean A, Lim H. Short-term outcomes in patients attending a primary care-based addiction shared care program. Can Fam Physician. 2009 Nov;55(11):1108-1109.e5. PMID 19910601
- [Background] Estee S, Wickizer T, He L, Shah MF, Mancuso D. Evaluation of the Washington state screening, brief intervention, and referral to treatment project: cost outcomes for Medicaid patients screened in hospital emergency departments. Med Care. 2010 Jan;48(1):18-24. doi: 10.1097/MLR.0b013e3181bd498f. PMID 19927016
- [Background] Fleming MF, Wilk A, Kruger J, Kropp S, Manwell L, Desnoyers P. Hospital-based alcohol and drug specialty consultation service: does it work? South Med J. 1995 Mar;88(3):275-82. doi: 10.1097/00007611-199503000-00006. PMID 7886522
- [Background] Friedmann PD, Hendrickson JC, Gerstein DR, Zhang Z, Stein MD. Do mechanisms that link addiction treatment patients to primary care influence subsequent utilization of emergency and hospital care? Med Care. 2006 Jan;44(1):8-15. doi: 10.1097/01.mlr.0000188913.50489.77. PMID 16365607
- [Background] McQueen J, Howe TE, Allan L, Mains D. Brief interventions for heavy alcohol users admitted to general hospital wards. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD005191. doi: 10.1002/14651858.CD005191.pub2. PMID 19588369
- [Background] Kahan M, Borgundvaag B, Midmer D, Borsoi D, Edwards C, Ladhani N. Treatment variability and outcome differences in the emergency department management of alcohol withdrawal. CJEM. 2005 Mar;7(2):87-92. doi: 10.1017/s1481803500013038. PMID 17355657
- [Background] Gray S, Borgundvaag B, Sirvastava A, Randall I, Kahan M. Feasibility and reliability of the SHOT: A short scale for measuring pretreatment severity of alcohol withdrawal in the emergency department. Acad Emerg Med. 2010 Oct;17(10):1048-54. doi: 10.1111/j.1553-2712.2010.00885.x. PMID 21040105
- [Background] Rumpf HJ, Hapke U, Meyer C, John U. Motivation to change drinking behavior: comparison of alcohol-dependent individuals in a general hospital and a general population sample. Gen Hosp Psychiatry. 1999 Sep-Oct;21(5):348-53. doi: 10.1016/s0163-8343(99)00032-8. PMID 10572776
- [Background] Solanki, D. R., D. Koyyalagunta, R. V. Shah, S. M. Silverman and L. Manchikanti (2011).
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Medications for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):505-14. doi: 10.7326/0003-4819-147-7-200710020-00008. PMID 17909211
- [Derived] Srivastava A, Clarke S, Hardy K, Kahan M. Facilitating rapid access to addiction treatment: a randomized controlled trial. Addict Sci Clin Pract. 2021 May 25;16(1):34. doi: 10.1186/s13722-021-00240-y. PMID 34034821